CLINICAL TRIAL: NCT05860400
Title: Efficacy and Safety of Comprehensive Treatment in Patients With Inflammation-associated Rapidly-progressive Coronary Artery Disease (IR-CAD): a Self-controlled Cohort Study
Brief Title: Efficacy and Safety of Comprehensive Treatment in Patients With IR-CAD: a Self-controlled Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, LiuZhenyu, Professor, Peking Union Medical College Hospital
Other Study IDs: K3483
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease; Coronary Artery Stenosis; Coronary Artery Restenosis; Coronary Artery Disease Progression; Inflammation; Inflammatory Disease; Inflammation Vascular
Keywords: Coronary Artery Disease; Coronary Revascularization; Progression, Disease; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Restenosis; Inflammation; Disease Progression | interventions — Secondary Prevention; Immunosuppression Therapy; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood samples will be retained for potential RNA sequencing, proteomics, and metabolomics studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-treatment Group: IR-CAD patients before receiving comprehensive treatment.
  Interventions: Behavioral: Healthy life style; Drug: Secondary prevention for atherosclerotic coronary artery disease; Procedure: Coronary revascularization; Drug: Supportive therapies
- Post-treatment Group: IR-CAD patients after receiving comprehensive treatment.
  Interventions: Behavioral: Healthy life style; Drug: Secondary prevention for atherosclerotic coronary artery disease; Drug: Immunosuppressive therapy; Procedure: Coronary revascularization; Drug: Supportive therapies

INTERVENTIONS:
Behavioral: Healthy life style — Healthy diet, regular exercise, and quitting smoking
Drug: Secondary prevention for atherosclerotic coronary artery disease — Antiplatelet therapy, as well as medications for control of heart rate, blood pressure, low-density lipoprotein cholesterol, and blood glucose
Drug: Immunosuppressive therapy — Glucocorticoids and/or immunosuppressive agents
  Groups: Post-treatment Group
Procedure: Coronary revascularization — Percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG).
Drug: Supportive therapies — Medical interventions for prevention and treatment of the side effects of the above treatment, such as abnormal liver function, hypocalcemia, hypokalemia, peptic ulcer, infection, et al.

SUMMARY:
This is a self-controlled cohort study to evaluate the efficacy and safety of comprehensive treatment in patients with inflammation-associated rapidly-progressive coronary artery disease (IR-CAD) by comparing the study endpoints before treatment with those after treatment in the same group of patients.

DETAILED DESCRIPTION:
A special type of coronary artery disease (CAD) has been identified in our clinical practice, which has completely different clinical features from those of typical atherosclerotic coronary artery disease (AS-CAD). The patients often have sterile inflammatory diseases and/or clinical evidence of inflammation, whose CAD progresses rapidly, recurs frequently, and responds poorly to intensified secondary prevention of AS-CAD, especially after percutaneous coronary intervention (PCI). We name this special type of CAD inflammation-associated rapidly-progressive coronary artery disease (IR-CAD).

The optimal treatment for IR-CAD remains unknown. We hypothesize that the rapid progression of IR-CAD might be associated with inflammation considering that: 1) inflammation is associated with poor prognosis in CAD patients after PCI; 2) IR-CAD patients often have sterile inflammatory diseases and/or clinical evidence of inflammation; 3) the disease progression of IR-CAD can be controlled to some extent with corticosteroids and immunosuppressive agents. Therefore, we incorporate immunosuppressive therapy into the overall management strategy of IR-CAD patients in clinical practice, developing comprehensive treatment, including: 1) intensified secondary prevention of AS-CAD; 2) immunosuppressive therapy; 3) coronary revascularization; 4) supportive therapies.

The present self-controlled cohort study is designed to evaluate the efficacy and safety of comprehensive treatment in about 39 IR-CAD patients by comparing the outcomes before with those after the initiation of comprehensive treatment in the same group of patients.

All patients who were admitted to the Department of Cardiology, Peking Union Medical College Hospital on and after January 1, 2022 will be screened for study participation. Patients were diagnosed as IR-CAD if they presented with 1) rapidly progressive myocardial ischemia (typical symptoms and non-invasive evidence) despite standard treatment for secondary prevention of AS-CAD after the last coronary revascularization; 2) angiographic evidence of new coronary lesions (de novo stenosis or restenosis) related to myocardial ischemia; 3) evidence of inflammation (positive inflammation markers or established diagnoses of inflammatory diseases or use of immunosuppressive therapy). IR-CAD patients who have received comprehensive treatment will be enrolled in the present cohort study. The eligible patients will be followed for 24 months since the initiation of comprehensive treatment.

The primary efficacy endpoint is major adverse cardiovascular events (MACE). The key secondary efficacy endpoint is target vessel related major adverse cardiovascular events (TV-MACE). Other secondary efficacy endpoints include individual components of MACE and TV-MACE, exercise capacity, angiographic metrics of coronary lesions, and inflammation markers. The safety endpoints are major bleeding events and severe infection events.

For endpoints which are categorical variables, e.g., MACE, survival analysis will be used to compare the survival curves before treatment (from the last coronary revascularization before the initiation of comprehensive treatment to the first occurrence of MACE) with those after treatment (from the initiation of comprehensive treatment to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first). Event-free survival rates and relative risk will be calculated.

For endpoints which are continuous variables, e.g., inflammation markers, paired t-test or paired rank sum test will be used to compare the endpoint levels before treatment (before the initiation of comprehensive treatment or at baseline) with those after treatment (the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, after the initiation of comprehensive treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling all the following criteria before initiation of comprehensive treatment:

   1.1 18 years of age or older, male or female.

   1.2 Negative result of urine or blood pregnancy test for females with childbearing potential (not post-menopausal or surgically sterile).

   1.3 Prior history of coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass graft [CABG]).

   1.4 Receiving standard treatment for secondary prevention of atherosclerotic coronary artery disease (AS-CAD) after the last coronary revascularization.

   1.5 Hospitalization due to rapidly-progressive myocardial ischemia:
   * Typical symptoms of angina (Canadian Cardiovascular Society [CCS] III-IV) and non-invasive evidence of myocardial ischemia; and
   * Occurred within 6 months or occurred on immunosuppressive therapy within 12 months of the last coronary revascularization.

   1.6 Angiographic evidence of new coronary lesions (de novo stenoses or restenoses):
   * Occurred after the last coronary revascularization; and
   * Related to myocardial ischemia (location, extent, severity, et al).

   1.7 Evidence of inflammation:
   * At least one of the markers indicating active inflammation has ever been elevated (erythrocyte sedimentation rate [ESR], high-sensitivity C-reactive protein [hs-CRP], interleukin [IL]-6, tumor necrosis factor [TNF]-α, ferritin, et al); or
   * Established diagnosis of systemic autoimmune disease or systemic vasculitis; or
   * Receiving immunosuppressive therapy.
2. Receiving comprehensive treatment, including ischemia-driven PCI which was performed no earlier than 40 days of the initiation of immunosuppressive therapy.

Exclusion Criteria:

1. Coronary restenosis due to mechanical factors (stent under-expansion, stent mal-apposition, stent rupture, et al).
2. Other moderate to severe heart diseases (congenital heart disease, valvular heart disease, myocarditis, cardiomyopathy, pericardial diseases, pulmonary hypertension, heart failure, arrhythmia, et al).
3. Active acute or chronic infection (human immunodeficiency virus [HIV], tuberculosis, et al).
4. Active malignancy (diagnosed within 12 months or with ongoing requirement for treatment).
5. Vital organ failure.
6. Life expectancy < 1 year.
7. Contraindications for or intolerance to treatment for secondary prevention of AS-CAD, contrast agents, glucocorticoids, immunosuppressive agents.
8. In pregnancy or breast-feeding, or with intention to be pregnant during the study period.
9. Risk of non-compliance (history of drug addiction or alcohol abuse, et al).
10. Previous enrollment in this study.
11. Participation in another study within 30 days.
12. Involvement in the planning and conduct of this study (applying to investigators, contract research organization staffs, study site staffs, et al).
13. Any condition, which in the opinion of the investigators, would make it unsuitable for the patient to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were admitted to the Department of Cardiology, Peking Union Medical College Hospital on and after January 1, 2022 will be screened for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  The composite endpoint including death, or Q wave myocardial infarction, or unplanned myocardial ischemia-driven coronary revascularization (PCI or CABG), or unplanned myocardial ischemia-driven hospitalization.

SECONDARY OUTCOMES:
Target vessel related major adverse cardiovascular events (TV-MACE) | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  The composite endpoint including cardiovascular death, or target vessel related Q wave myocardial infarction, or target vessel related unplanned myocardial ischemia-driven coronary revascularization (PCI or CABG), or target vessel related unplanned myocardial ischemia-driven hospitalization.
Death | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  All-cause death.
Myocardial infarction | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Myocardial injury due to myocardial ischemia.
Target vessel related myocardial infarction | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Myocardial infarction in the area supplied by the target vessel.
Unplanned myocardial ischemia-driven coronary revascularization | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Unplanned coronary revascularization (PCI or CABG) due to myocardial ischemia.
Target vessel related unplanned myocardial ischemia-driven coronary revascularization | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Unplanned coronary revascularization (PCI or CABG) in the target vessel due to myocardial ischemia.
Unplanned myocardial ischemia-driven hospitalization | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Unplanned hospitalization due to myocardial ischemia.
Target vessel related unplanned myocardial ischemia-driven hospitalization | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Unplanned hospitalization due to myocardial ischemia in the area supplied by the target vessel.
Walking distance in 6 minutes | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of 6-minute walk test (6MWT).
Number of squats in 1 minute | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of 1-minute squatting test (1MST).
Target lesion minimal lumen area (TL-MLA) | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The minimum lumen area of the target lesion on optical coherence tomography (OCT).
Target lesion percent area stenosis (TL-%AS) | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  Percent area stenosis (% AS) = { [ ( proximal RLA + distal RLA ) - (MLA × 2) ] / ( proximal RLA + distal RLA ) } × 100% in the cross-section with the MLA of the target lesion on optical coherence tomography (OCT). RLA = reference lumen area; MLA = minimum lumen area; % AS = percent area stenosis.
SYNTAX score | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of SYNTAX score calculation.
Number of vessel segments with coronary lesions | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  Number of vessel segments with diameter stenosis ≥ 50% on coronary angiogram.
Erythrocyte sedimentation rate (ESR) | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of erythrocyte sedimentation rate (ESR) test.
High-sensitivity C-reactive protein (hs-CRP) | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of serum high-sensitivity C-reactive protein (hs-CRP) test.
interleukin (IL)-6 | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of serum interleukin (IL)-6 test.
Tumor necrosis factor (TNF)-α | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of serum tumor necrosis factor (TNF)-α test.
Birmingham vasculitis activity score | Before treatment: the timepoint before the initiation of comprehensive treatment, or at baseline. After treatment: the timepoint of the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first.
  The result of Birmingham Vasculitis Activity Score (version 3) calculation.

OTHER OUTCOMES:
Major bleeding events | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Major bleeding events evaluated according to the Bleeding Academic Research Consortium (BARC) criteria.
Severe infection events | Time from the last coronary revascularization to the first occurrence of MACE, or the last follow-up visit, or the end of 24-month follow-up, which occurs first, both before and after the initiation of comprehensive treatment.
  Infection events involving vital organs, or with complications (such as structural change and/or dysfunction of vital organs, septic shock), or requiring hospitalization, or requiring treatment with intravenous antibiotics, or requiring treatment with interventional procedures or surgeries.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liu, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Neumann FJ, Sousa-Uva M. 'Ten commandments' for the 2018 ESC/EACTS Guidelines on Myocardial Revascularization. Eur Heart J. 2019 Jan 7;40(2):79-80. doi: 10.1093/eurheartj/ehy855. No abstract available. PMID 30615155
- [Background] Fernandez DM, Giannarelli C. Immune cell profiling in atherosclerosis: role in research and precision medicine. Nat Rev Cardiol. 2022 Jan;19(1):43-58. doi: 10.1038/s41569-021-00589-2. Epub 2021 Jul 15. PMID 34267377
- [Background] Deroissart J, Porsch F, Koller T, Binder CJ. Anti-inflammatory and Immunomodulatory Therapies in Atherosclerosis. Handb Exp Pharmacol. 2022;270:359-404. doi: 10.1007/164_2021_505. PMID 34251531
- [Background] Engelen SE, Robinson AJB, Zurke YX, Monaco C. Therapeutic strategies targeting inflammation and immunity in atherosclerosis: how to proceed? Nat Rev Cardiol. 2022 Aug;19(8):522-542. doi: 10.1038/s41569-021-00668-4. Epub 2022 Jan 31. PMID 35102320
- [Background] Tucker B, Vaidya K, Cochran BJ, Patel S. Inflammation during Percutaneous Coronary Intervention-Prognostic Value, Mechanisms and Therapeutic Targets. Cells. 2021 Jun 4;10(6):1391. doi: 10.3390/cells10061391. PMID 34199975
- [Background] Kalkman DN, Aquino M, Claessen BE, Baber U, Guedeney P, Sorrentino S, Vogel B, de Winter RJ, Sweeny J, Kovacic JC, Shah S, Vijay P, Barman N, Kini A, Sharma S, Dangas GD, Mehran R. Residual inflammatory risk and the impact on clinical outcomes in patients after percutaneous coronary interventions. Eur Heart J. 2018 Dec 7;39(46):4101-4108. doi: 10.1093/eurheartj/ehy633. PMID 30358832
- [Background] Guedeney P, Claessen BE, Kalkman DN, Aquino M, Sorrentino S, Giustino G, Farhan S, Vogel B, Sartori S, Montalescot G, Sweeny J, Kovacic JC, Krishnan P, Barman N, Dangas G, Kini A, Baber U, Sharma S, Mehran R. Residual Inflammatory Risk in Patients With Low LDL Cholesterol Levels Undergoing Percutaneous Coronary Intervention. J Am Coll Cardiol. 2019 May 21;73(19):2401-2409. doi: 10.1016/j.jacc.2019.01.077. PMID 31097159
- [Background] Takahashi N, Dohi T, Endo H, Funamizu T, Wada H, Doi S, Kato Y, Ogita M, Okai I, Iwata H, Okazaki S, Isoda K, Miyauchi K, Shimada K. Residual Inflammation Indicated by High-Sensitivity C-Reactive Protein Predicts Worse Long-Term Clinical Outcomes in Japanese Patients after Percutaneous Coronary Intervention. J Clin Med. 2020 Apr 6;9(4):1033. doi: 10.3390/jcm9041033. PMID 32268533
- [Background] Kikuchi S, Okada K, Hibi K, Maejima N, Yabu N, Uchida K, Tamura K, Kimura K. Coronary arteritis: a case series. Eur Heart J Case Rep. 2020 Feb 17;4(2):1-6. doi: 10.1093/ehjcr/ytaa011. eCollection 2020 Apr. PMID 32352046
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; ESC Scientific Document Group. Fourth universal definition of myocardial infarction (2018). Eur Heart J. 2019 Jan 14;40(3):237-269. doi: 10.1093/eurheartj/ehy462. No abstract available. PMID 30165617
- [Background] Braunwald E. Unstable angina. A classification. Circulation. 1989 Aug;80(2):410-4. doi: 10.1161/01.cir.80.2.410. No abstract available. PMID 2752565
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242